CLINICAL TRIAL: NCT04535167
Title: A PHASE 1B, 2-PART, DOUBLE-BLIND, PLACEBO-CONTROLLED, SPONSOR-OPEN STUDY, TO EVALUATE THE SAFETY, TOLERABILITY AND PHARMACOKINETICS OF SINGLE ASCENDING (24-HOUR, PART 1) AND MULTIPLE ASCENDING (120-HOUR, PART 2) INTRAVENOUS INFUSIONS OF PF-07304814 IN HOSPITALIZED PARTICIPANTS WITH COVID-19
Brief Title: First-In-Human Study To Evaluate Safety, Tolerability, And Pharmacokinetics Following Single Ascending And Multiple Ascending Doses of PF-07304814 In Hospitalized Participants With COVID-19.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: C4611001; 2020-003905-73 (EudraCT Number)
Record Dates: First submitted 2020-08-21; First posted 2020-09-01 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Viral Disease
Keywords: COVID-19; SARS-COV-2
MeSH Terms: conditions — Virus Diseases; COVID-19 | interventions — lufotrelvir

STUDY DESIGN:
Intervention Model Description: Part 1 will have 2 planned cohorts. Each escalating cohort will be initiated for enrollment after assessment of safety, tolerability and PK data from previous cohorts by an independent IRC and is deemed acceptable.
  Part 2 will have 2 planned cohort and each escalating cohort will be initiated after all safety, tolerability and PK data from previous cohort is evaluated and is deemed acceptable by a competent regulatory authority.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-07304814 (Experimental): Part 1:
  Cohort 1-5
  Part 2:
  Cohort 6-9
  Interventions: Drug: PF-07304814
- Placebo (Placebo Comparator): Part 1:
  Cohort 1-5
  Part 2:
  Cohort 6-9
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-07304814 — PF-07304814 is an anti-viral, formulated for intravenous delivery
  Arms: PF-07304814
Drug: Placebo — Placebo will be formulated for intravenous delivery
  Arms: Placebo

SUMMARY:
It is Phase 1b, 2-part, double-blind, placebo-controlled study to evaluate safety, tolerability, and pharmacokinetics of PF-07304814, in patients hospitalized with SARS-CoV-2 virus infection.

DETAILED DESCRIPTION:
It is a 2-part study in hospitalized COVID-19 patients.

* Part 1 is to evaluate safety, tolerability, PK and markers of clinical activity of escalating doses of PF-07304814 given as 24-hour IV infusion.

  2 planned and 3 optional cohorts with 8 participants each are planned.
* Part 2 is to evaluate safety, tolerability, PK and markers of clinical activity of escalating doses of PF- 07304814 given as 120-hour infusion.

  2 planned and 2 optional cohorts with 8 participants each are planned

ELIGIBILITY:
* Inclusion Criteria:

  1. Male or female participants between the ages of 18 and 79 years.
  2. Confirmed SARS-CoV-2 infection.
  3. Hospitalized for COVID-19.
  4. Symptoms consistent with COVID-19 indicated by at least 1 of the following: fever, cough, sore throat, malaise, headache, muscle pain, shortness of breath, new loss of taste and smell, nausea, chills, fatigue, rhinorrhea, diarrhea, vomiting or radiographic infiltrates by imaging consistent with COVID-19
  5. Total body weight >=50 kg (110 lb), BMI <40 kg/m2; BMI <35 kg/m2 for 76- 79 years.
* Exclusion Criteria:

  1. Evidence of critical illness, defined by at least one of the following: Respiratory failure, Multi-organ dysfunction/failure, Cardiac failure or septic shock
  2. Participants that are anticipated by the study Investigator to progress to critical disease, including mechanical ventilation, within 24 hours of enrolment
  3. Participants with pre-existing moderate to severe cardiovascular disease, uncontrolled diabetes, or severe asthma or severe COPD.

  3.Participants with a known medical history of recent acute or chronic liver disease (other than NASH), chronic or active hepatitis B or C infection, or primary biliary cirrhosis.

  4.Participants with a known medical history of ischemic heart disease, heart failure, dysrhythmia or other pre-existing cardiac condition.

  5. Participants with known HIV infection, acute or chronic history of hepatitis B or C.

  6.Participants with a known medical history of recurrent seizures. 7. Participants with history of venous thromboembolic event, including deep venous thrombosis or pulmonary embolism 8.Confirmed concurrent active systemic infection other than COVID-19. 9.Current diagnosis of cancer, unless in remission and untreated. 10.Other medical or psychiatric condition including recent or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation 11.Females who are pregnant or breastfeeding.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- United States (9):
  - El Camino Health, Mountain View, California
  - Palo Alto Medical Foundation, Mountain View, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - UC Davis Health Investigational Drug Pharmacy, Sacramento, California
  - UC Davis Medical Center, Sacramento, California
  - Massachusetts General Hospital Translational and Clinical Research Center, Boston, Massachusetts
  - Massachusetts General Hospital, Clinical Trials Pharmacy, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Regional One Health, Memphis, Tennessee
- University Hospital Brugmann, Brussels, Belgium
- Santa Casa De Misericórdia de Belo Horizonte, Belo Horizonte, Minas Gerais, Brazil
- Spain (2):
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Virgen Del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Robinson P, Toussi SS, Aggarwal S, Bergman A, Zhu T, Hackman F, Sathish JG, Updyke L, Loudon P, Krishna G, Clevenbergh P, Hernandez-Mora MG, Cisneros Herreros JM, Albertson TE, Dougan M, Thacker A, Baniecki ML, Soares H, Whitlock M, Nucci G, Menon S, Anderson AS, Binks M. Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Intravenous Infusions of PF-07304814 (Lufotrelvir) in Participants Hospitalized With COVID-19. Open Forum Infect Dis. 2023 Jul 10;10(8):ofad355. doi: 10.1093/ofid/ofad355. eCollection 2023 Aug. PMID 37559753
- [Derived] Crosas-Molist E, Samain R, Kohlhammer L, Orgaz JL, George SL, Maiques O, Barcelo J, Sanz-Moreno V. Rho GTPase signaling in cancer progression and dissemination. Physiol Rev. 2022 Jan 1;102(1):455-510. doi: 10.1152/physrev.00045.2020. Epub 2021 Sep 20. PMID 34541899
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4611001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 26 hospitalized participants with COVID-19 were enrolled in this study. 25 participants were randomized to receive single ascending (24-hour, part 1) or multiple ascending (120-hour, part 2) intravenous infusions of PF-07304814 or placebo. One participant was not treated and discontinued from study due to being incorrectly randomized. All reported data are on 25 participants who were randomized and received at least 1 dose of PF-07304814 or placebo (referred to as "enrolled" herein).
Groups:
- Part 1: PF-07304814 500 mg 24-hours Continuous Infusion: Participants were enrolled in this arm and received PF-07304814 500 mg as 24-hour continuous intravenous infusion.
- Part 1: PF-07304814 250 mg 24-hours Continuous Infusion: Participants were enrolled in this arm and received PF-07304814 250 mg as 24-hour continuous intravenous infusion.
- Part 1: 500 mg Placebo 24-hours Continuous Infusion; Part 1: 250 mg Placebo 24-hours Continuous Infusion: Participants were enrolled in this arm and received placebo as 24-hour continuous intravenous infusion.
- Part 2: PF-07304814 500 mg 120-hours Continuous Infusion: Participants were enrolled in this arm and received PF-07304814 500 mg daily as 5-day (~120 hours) continuous intravenous infusion.
- Part 2: PF-07304814 250 mg 120-hours Continuous Infusion: Participants were enrolled in this arm and received PF-07304814 250 mg daily as 5-day (~120 hours) continuous intravenous infusion.
- Part 2: Placebo 120-hours Continuous Infusion: Participants were enrolled in this arm and received placebo as 5-day (~120 hours) continuous intravenous infusion.
Period: Treatment
Arm/Group | Part 1: PF-07304814 500 mg 24-hours Continuous Infusion | Part 1: PF-07304814 250 mg 24-hours Continuous Infusion | Part 1: 500 mg Placebo 24-hours Continuous Infusion | Part 1: 250 mg Placebo 24-hours Continuous Infusion | Part 2: PF-07304814 500 mg 120-hours Continuous Infusion | Part 2: PF-07304814 250 mg 120-hours Continuous Infusion | Part 2: Placebo 120-hours Continuous Infusion
Started | 2 | 2 | 2 | 2 | 6 | 7 | 4
Completed | 2 | 2 | 2 | 2 | 6 | 7 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Follow-Up
Arm/Group | Part 1: PF-07304814 500 mg 24-hours Continuous Infusion | Part 1: PF-07304814 250 mg 24-hours Continuous Infusion | Part 1: 500 mg Placebo 24-hours Continuous Infusion | Part 1: 250 mg Placebo 24-hours Continuous Infusion | Part 2: PF-07304814 500 mg 120-hours Continuous Infusion | Part 2: PF-07304814 250 mg 120-hours Continuous Infusion | Part 2: Placebo 120-hours Continuous Infusion
Started | 2 | 2 | 2 | 2 | 6 | 7 | 4 (Participant may or may not continued in follow-up period after discontinuing from the treatment period.)
Completed | 2 | 2 | 2 | 1 | 6 | 7 | 3
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: PF-07304814 500 mg 24-hours Continuous Infusion | Part 1: PF-07304814 250 mg 24-hours Continuous Infusion | Part 1: 500 mg Placebo 24-hours Continuous Infusion | Part 1: 250 mg Placebo 24-hours Continuous Infusion | Part 2: PF-07304814 500 mg 120-hours Continuous Infusion | Part 2: PF-07304814 250 mg 120-hours Continuous Infusion | Part 2: Placebo 120-hours Continuous Infusion | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 6 | 7 | 4 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 2 | 1 | 5 | 5 | 2 | 18
  >=65 years | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 6
  Male | 1 | 2 | 1 | 1 | 4 | 6 | 4 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 4
  Not Hispanic or Latino | 1 | 2 | 1 | 2 | 4 | 5 | 3 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
  White | 2 | 1 | 1 | 2 | 5 | 5 | 3 | 19
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With TEAEs, SAEs, and Severe TEAEs - Part 1: SAD
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious adverse event (SAE) was defined as an AE: 1. resulting in death, 2. was life-threatening, 3. required inpatient hospitalization or prolongation of existing hospitalization, 4. resulted in persistent disability, 5. was a congenital anomaly/birth defect, or considered to be an important medical event. An adverse event was considered a Treatment-Emergent Adverse Event (TEAE) if the event started during the effective duration of treatment.
Time Frame: Day 1 to 37 days
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention for the given part of the study (Part 1: SAD). Participants were analyzed according to the product they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-07304814 500 mg 24-hours Continuous Infusion | Part 1: PF-07304814 250 mg 24-hours Continuous Infusion | Part 1: 500 mg Placebo 24-hours Continuous Infusion | Part 1: 250 mg Placebo 24-hours Continuous Infusion
Number analyzed (Participants) | 2 | 2 | 2 | 2
Participants
  All-causality TEAEs | 1 | 1 | 2 | 2
  Treatment-related TEAEs | 0 | 0 | 1 | 1
  All-causality SAEs | 1 | 0 | 1 | 1
  Treatment-related SAEs | 0 | 0 | 0 | 0
  All-causality severe AEs | 1 | 1 | 1 | 1
  Treatment-related severe AEs | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With TEAEs, SAEs, and Severe TEAEs - Part 2: MAD
Description: as for outcome 1
Time Frame: Day 1 to 41 days
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention for the given part of the study (Part 2: MAD). Participants were analyzed according to the product they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: PF-07304814 500 mg 120-hours Continuous Infusion | Part 2: PF-07304814 250 mg 120-hours Continuous Infusion | Part 2: Placebo 120-hours Continuous Infusion
Number analyzed (Participants) | 6 | 7 | 4
Participants
  All-causality TEAEs | 2 | 4 | 3
  Treatment-related TEAEs | 0 | 0 | 1
  All-causality SAEs | 1 | 2 | 1
  Treatment-related SAEs | 0 | 0 | 0
  All-causality severe AEs | 0 | 2 | 1
  Treatment-related severe AEs | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Discontinuations From Study/Study Drug or Dose Reduction Due to TEAEs - Part 1: SAD
Description: An AE was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE was considered a TEAE if the event started during the effective duration of treatment.
Time Frame: Day 1 up to 37 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-07304814 500 mg 24-hours Continuous Infusion | Part 1: PF-07304814 250 mg 24-hours Continuous Infusion | Part 1: 500 mg Placebo 24-hours Continuous Infusion | Part 1: 250 mg Placebo 24-hours Continuous Infusion
Number analyzed (Participants) | 2 | 2 | 2 | 2
Participants
  Discontinued from study due to adverse events | 0 | 0 | 0 | 0
  Discontinuation from study drug due to AE and continued study | 0 | 0 | 0 | 0
  Dose reduced or temporary discontinuation due to adverse events | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Discontinuations From Study/Study Drug or Dose Reduction Due to TEAEs - Part 2: MAD
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE was considered a Treatment-Emergent Adverse Event (TEAE) if the event started during the effective duration of treatment.
Time Frame: Day 1 to 41 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: PF-07304814 500 mg 120-hours Continuous Infusion | Part 2: PF-07304814 250 mg 120-hours Continuous Infusion | Part 2: Placebo 120-hours Continuous Infusion
Number analyzed (Participants) | 6 | 7 | 4
Participants
  Discontinued from study due to adverse events | 0 | 0 | 1
  Discontinuation from study drug due to AE and continued study | 0 | 0 | 0
  Dose reduced or temporary discontinuation due to adverse events | 1 | 0 | 0

5. Primary Outcome: Number of Participants With Laboratory Abnormality Without Regard to Baseline Abnormality - Part 1: SAD
Description: Laboratory abnormalities reported in at least 1 participant are presented in this OM, including: Hematology - lymphocytes, basophiles; Clinical Chemistry - aspartate aminotransferase, alanine aminotransferase, calcium, bicarbonate, glucose, glucose -FASTING; Urinalysis - urine glucose, urine hemoglobin, urobilinogen and urine erythrocytes (per high power field).
  Baseline was the last pre-dose measurement. LLN = lower limit of normal, ULN = upper limit of normal.
Time Frame: Day 1 up to 6 days
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention for the given part of the study (Part 1: SAD). Participants were analyzed according to the product they actually received.
  Number of Participants analyzed refers to number of participants evaluable for this OM; Number Analyzed refers to number of participants evaluable at the specific parameters.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-07304814 500 mg 24-hours Continuous Infusion | Part 1: PF-07304814 250 mg 24-hours Continuous Infusion | Part 1: 500 mg Placebo 24-hours Continuous Infusion | Part 1: 250 mg Placebo 24-hours Continuous Infusion
Number analyzed (Participants) | 2 | 2 | 2 | 2
Participants
  Lymphocytes (10^3/mm3) < 0.8*LLN | 1 | 2 | 0 | 1
  Basophils (10^3/mm3) > 1.2*ULN | 0 | 0 | 1 | 0
  Aspartate Aminotransferase (U/L) > 3.0*ULN | 0 | 1 | 0 | 1
  Alanine Aminotransferase (U/L) > 3.0*ULN | 0 | 1 | 1 | 0
  Calcium (mg/dL) < 0.9*LLN | 0 | 0 | 1 | 0
  Bicarbonate (mEq/L) < 0.9*LLN | 0 | 1 | 1 | 1
  Glucose (mg/dL) > 1.5*ULN: number analyzed (Participants) | 0 | 2 | 0 | 2
  Glucose (mg/dL) > 1.5*ULN | 0 | 1 | 0 | 2
  Glucose - FASTING (mg/dL) >1.5*ULN: number analyzed (Participants) | 2 | 0 | 2 | 0
  Glucose - FASTING (mg/dL) >1.5*ULN | 1 | 0 | 2 | 0
  URINE Glucose ≥ 1 | 1 | 0 | 0 | 0
  URINE Hemoglobin ≥ 1 | 0 | 0 | 0 | 1
  Urobilinogen ≥ 1 | 0 | 0 | 0 | 1
  URINE Erythrocytes (/HPF) ≥ 20: number analyzed (Participants) | 0 | 1 | 1 | 2
  URINE Erythrocytes (/HPF) ≥ 20 | 0 | 0 | 0 | 1

6. Primary Outcome: Number of Participants With Laboratory Abnormality Without Regard to Baseline Abnormality - Part 2: MAD
Description: Laboratory abnormalities reported in at least 1 participant are presented in this OM, including: Hematology - lymphocytes hemoglobin, hematocrit, erythrocytes, ery. mean corpuscular volume, ery. mean corpuscular, hemoglobin; Clinical Chemistry - alanine aminotransferase, protein, albumin, urea nitrogen, creatinine, HDL cholesterol, triglycerides, calcium, phosphate, bicarbonate, glucose; Urinalysis - urine glucose, ketones, urine hemoglobin, urobilinogen, nitrite, leukocyte esterase, urine erythrocytes (per high power field), urine leukocytes (Scalar).
  Baseline was the last pre-dose measurement. LLN = lower limit of normal, ULN = upper limit of normal
Time Frame: Day 1 up to 41 days
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention for the given part of the study (Part 2: MAD). Participants were analyzed according to the product they actually received.
  Number of Participants analyzed refers to number of participants evaluable for this OM; Number Analyzed refers to number of participants evaluable at the specific parameters.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: PF-07304814 500 mg 120-hours Continuous Infusion | Part 2: PF-07304814 250 mg 120-hours Continuous Infusion | Part 2: Placebo 120-hours Continuous Infusion
Number analyzed (Participants) | 6 | 7 | 4
Participants
  Hemoglobin (g/dL)<0.8*LLN | 0 | 2 | 1
  Hematocrit (%)<0.8x LLN | 0 | 2 | 0
  Erythrocytes (10^6/mm3)<0.8x LLN | 0 | 1 | 0
  Ery. mean corpuscular volume (um^3)<0.9*LLN | 0 | 1 | 1
  Ery. mean corpuscular hemoglobin (pg/cell)<0.9*LLN | 0 | 1 | 1
  Lymphocytes (10^3/mm3)<0.8x LLN | 0 | 3 | 3
  Alanine aminotransferase (U/L)>3.0*ULN | 0 | 1 | 1
  Protein (g/dL)<0.8x LLN | 0 | 1 | 1
  Albumin (g/dL) <0.8x LLN | 1 | 0 | 1
  Urea nitrogen (mg/dL)>1.3x ULN | 0 | 0 | 1
  Creatinine (mg/dL)>1.3x ULN | 0 | 0 | 1
  HDL cholesterol (mg/dL)<0.8x LLN | 2 | 3 | 1
  Triglycerides (mg/dL)>1.3x ULN | 1 | 1 | 0
  Calcium (mg/dL)<0.9x LLN | 1 | 1 | 0
  Phosphate (mg/dL)<0.8x LLN | 0 | 1 | 0
  Bicarbonate (mEq/L)<0.9x LLN | 2 | 4 | 3
  Glucose (mg/dL)>1.5x ULN | 3 | 6 | 2
  URINE glucose≥1 | 1 | 1 | 0
  Ketones≥1 | 0 | 1 | 0
  Urine hemoglobin ≥ 1 | 1 | 2 | 1
  Urobilinogen≥1 | 1 | 2 | 1
  Nitrite≥1 | 1 | 0 | 0
  Leukocyte esterase ≥ 1 | 1 | 2 | 0
  Urine erythrocytes (/HPF)≥20: number analyzed (Participants) | 5 | 5 | 3
  Urine erythrocytes (/HPF)≥20 | 1 | 2 | 0
  Urine leukocytes (Scalar)≥20: number analyzed (Participants) | 5 | 6 | 3
  Urine leukocytes (Scalar)≥20 | 0 | 1 | 0

7. Primary Outcome: Summary of Baseline and Change From Baseline in Systolic and Diastolic Blood Pressure at Day 1 (30 Minutes, 2 Hours, 6 Hour, and 12 Hours; 24 Hours [End of Treatment]), Day 3 (Follow-up 1) and Day 6 (Follow-up 2) - Part 1: SAD
Description: Absolute baseline values and changes from baseline in supine systolic and diastolic blood pressure were summarized by treatment and time post-dose. Blood pressure was assessed in the supine position after at least 5 minutes of rest in a quiet setting without distractions. Baseline was defined as the last pre-dose measurement.
Time Frame: Baseline (pre-dose Day 1), Day 1-30 minutes, 2 hours, 6 hour, and 12 hours; 24 hours (End of Treatment), Day 3 (Follow-up 1) and Day 6 (Follow-up 2).
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention for Part 1 (SAD) of the study. Participants were be analyzed according to the product they received.
  Number of Participants analyzed refers to number of participants evaluable for this OM; Number Analyzed refers to number of participants evaluable at the specific time point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part 1: PF-07304814 500 mg 24-hours Continuous Infusion | Part 1: PF-07304814 250 mg 24-hours Continuous Infusion | Part 1: 500 mg Placebo 24-hours Continuous Infusion | Part 1: 250 mg Placebo 24-hours Continuous Infusion
Number analyzed (Participants) | 2 | 2 | 2 | 2
mmHg
  Systolic blood pressure: Baseline | 116.0 (4.24) | 134.5 (13.44) | 108.0 (14.14) | 127.5 (30.41)
  Systolic blood pressure: Change from Baseline: Day 1- 30 minutes | 6.0 (18.38) | -12.5 (12.02) | -4.0 (12.73) | 9.5 (17.68)
  Systolic blood pressure: Change from Baseline: Day 1 - 2 hours | 12.0 (22.63) | -20.0 (11.31) | 4.0 (2.83) | 3.5 (20.51)
  Systolic blood pressure: Change from Baseline: Day 1 - 6 hours | -1.5 (14.85) | -20.5 (13.44) | 0.0 (7.07) | 16.5 (24.75)
  Systolic blood pressure: Change from Baseline: Day 1 - 12 hours | -8.0 (18.38) | -6.5 (26.16) | -2.5 (4.95) | 10.0 (5.66)
  Systolic blood pressure: Change from Baseline: End of Treatment: number analyzed (Participants) | 2 | 1 | 2 | 2
  Systolic blood pressure: Change from Baseline: End of Treatment | -5.0 (16.97) | -17.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 0.0 (8.49) | -1.0 (5.66)
  Systolic blood pressure: Change from Baseline: Follow Up 1 | 8.0 (11.31) | -16.5 (21.92) | -3.0 (9.90) | 13.5 (3.54)
  Systolic blood pressure: Change from Baseline: Follow Up 2: number analyzed (Participants) | 1 | 1 | 1 | 2
  Systolic blood pressure: Change from Baseline: Follow Up 2 | 17.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -20.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -6.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -14.5 (27.58)
  Diastolic blood pressure: Baseline | 64.0 (9.90) | 59.0 (21.21) | 68.5 (13.44) | 76.5 (9.19)
  Diastolic blood pressure: Change from Baseline: Day 1 - 30 minutes | 5.0 (5.66) | 16.0 (14.14) | -5.0 (8.49) | 6.0 (9.90)
  Diastolic blood pressure: Change from Baseline: Day 1 - 2 hours | 9.5 (12.02) | 11.5 (7.78) | -2.0 (4.24) | 3.0 (11.31)
  Diastolic blood pressure: Change from Baseline: Day 1 - 6 hours | -1.5 (6.36) | 8.5 (17.68) | -8.0 (7.07) | 6.5 (7.78)
  Diastolic blood pressure: Change from Baseline: Day 1 - 12 hours | 9.0 (9.90) | 13.0 (16.97) | -8.5 (2.12) | -1.0 (0.00)
  Diastolic blood pressure: Change from Baseline: End of Treatment: number analyzed (Participants) | 2 | 1 | 2 | 2
  Diastolic blood pressure: Change from Baseline: End of Treatment | -1.0 (0.00) | 23.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -7.5 (6.36) | -4.5 (0.71)
  Diastolic blood pressure: Change from Baseline: Follow Up 1 | 17.0 (2.83) | 6.0 (2.83) | -6.0 (1.41) | 8.5 (2.12)
  Diastolic blood pressure: Change from Baseline: Follow Up 2: number analyzed (Participants) | 1 | 1 | 1 | 2
  Diastolic blood pressure: Change from Baseline: Follow Up 2 | 12.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed | 17.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed | -11.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed | -2.0 (12.73)

8. Primary Outcome: Summary of Baseline and Change From Baseline in Systolic and Diastolic Blood Pressure at Day2,3,4,5, and 6 (120 Hours), Day7 (Follow-up 1), Day10 (Follow-up 2), Day14 (Follow-up 3), Between Day34-41 (Follow-up 4), and/or Early Termination - Part 2: MAD
Description: as for outcome 7
Time Frame: Baseline (pre-dose Day 1), Day 2, 3, 4, 5; 120 hours (End of Treatment), Day 7 (Follow-up 1), Day 10 (Follow-up 2), Day 14 (Follow-up 3), Follow-up 4 (between Day 34-41) and/or early termination (ET) .
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention for Part 2 (MAD) of the study. Participants were be analyzed according to the product they received.
  Number of Participants analyzed refers to number of participants evaluable for this OM; Number Analyzed refers to number of participants evaluable at the specific time point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part 2: PF-07304814 500 mg 120-hours Continuous Infusion | Part 2: PF-07304814 250 mg 120-hours Continuous Infusion | Part 2: Placebo 120-hours Continuous Infusion
Number analyzed (Participants) | 6 | 7 | 4
mmHg
  Systolic blood pressure: Baseline | 105.3 (18.08) | 127.6 (13.64) | 116.5 (14.29)
  Systolic blood pressure: Change from Baseline: Day 2 | 4.8 (10.34) | 1.4 (14.20) | -4.3 (8.42)
  Systolic blood pressure: Change from Baseline: Day 3 | 15.5 (14.15) | -4.9 (16.92) | 10.8 (24.70)
  Systolic blood pressure: Change from Baseline: Day 4: number analyzed (Participants) | 6 | 7 | 3
  Systolic blood pressure: Change from Baseline: Day 4 | -1.2 (12.54) | -13.1 (13.59) | -18.0 (6.00)
  Systolic blood pressure: Change from Baseline: Day 5: number analyzed (Participants) | 6 | 7 | 3
  Systolic blood pressure: Change from Baseline: Day 5 | 3.2 (10.28) | -4.6 (14.14) | -12.3 (6.66)
  Systolic blood pressure: Change from Baseline: End of Treatment: number analyzed (Participants) | 6 | 7 | 3
  Systolic blood pressure: Change from Baseline: End of Treatment | 3.7 (14.85) | -11.6 (12.71) | -11.0 (6.08)
  Systolic blood pressure: Change from Baseline: Early Termination: number analyzed (Participants) | 0 | 0 | 1
  Systolic blood pressure: Change from Baseline: Early Termination |  |  | 11.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  Systolic blood pressure: Change from Baseline: Follow Up 1 | 5.0 (14.14) | -7.7 (10.83) | 4.5 (17.29)
  Systolic blood pressure: Change from Baseline: Follow Up 2: number analyzed (Participants) | 4 | 1 | 2
  Systolic blood pressure: Change from Baseline: Follow Up 2 | 21.5 (17.62) | 1.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 24.0 (48.08)
  Systolic blood pressure: Change from Baseline: Follow Up 3: number analyzed (Participants) | 4 | 2 | 3
  Systolic blood pressure: Change from Baseline: Follow Up 3 | 19.0 (14.07) | -1.0 (2.83) | 11.7 (17.01)
  Systolic blood pressure: Change from Baseline: Follow Up 4: number analyzed (Participants) | 2 | 3 | 1
  Systolic blood pressure: Change from Baseline: Follow Up 4 | 15.0 (2.83) | -2.7 (6.66) | 15.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  Diastolic blood pressure: Baseline | 63.8 (11.39) | 78.7 (7.87) | 72.0 (12.52)
  Diastolic blood pressure: Change from Baseline: Day 2 | 4.7 (10.52) | -2.4 (7.48) | 1.0 (9.83)
  Diastolic blood pressure: Change from Baseline: Day 3 | 7.8 (10.96) | -9.4 (13.15) | 2.3 (9.54)
  Diastolic blood pressure: Change from Baseline: Day 4: number analyzed (Participants) | 6 | 7 | 3
  Diastolic blood pressure: Change from Baseline: Day 4 | 2.7 (8.57) | -7.4 (9.32) | -11.7 (4.93)
  Diastolic blood pressure: Change from Baseline: Day 5: number analyzed (Participants) | 6 | 7 | 3
  Diastolic blood pressure: Change from Baseline: Day 5 | 2.7 (10.05) | -9.6 (11.62) | 2.0 (11.27)
  Diastolic blood pressure: Change from Baseline: End of Treatment: number analyzed (Participants) | 6 | 7 | 3
  Diastolic blood pressure: Change from Baseline: End of Treatment | 2.5 (8.96) | -7.9 (17.00) | -13.0 (2.00)
  Diastolic blood pressure: Change from Baseline: Early Termination: number analyzed (Participants) | 0 | 0 | 1
  Diastolic blood pressure: Change from Baseline: Early Termination |  |  | 11.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  Diastolic blood pressure: Change from Baseline: Follow Up 1 | 4.8 (11.34) | -6.7 (13.86) | -5.8 (12.04)
  Diastolic blood pressure: Change from Baseline: Follow Up 2: number analyzed (Participants) | 4 | 1 | 2
  Diastolic blood pressure: Change from Baseline: Follow Up 2 | 15.5 (13.48) | -34.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -3.0 (1.41)
  Diastolic blood pressure: Change from Baseline: Follow Up 3: number analyzed (Participants) | 4 | 2 | 3
  Diastolic blood pressure: Change from Baseline: Follow Up 3 | 13.0 (13.64) | -14.5 (13.44) | 5.0 (21.63)
  Diastolic blood pressure: Change from Baseline: Follow Up 4: number analyzed (Participants) | 2 | 3 | 1
  Diastolic blood pressure: Change from Baseline: Follow Up 4 | 11.0 (14.14) | -4.3 (12.66) | 12.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.

9. Primary Outcome: Summary of Baseline and Change From Baseline in Pulse Rate at Day 1 (30 Minutes, 2 Hours, 6 Hour, and 12 Hours; 24 Hours [End of Treatment]), Day 3 (Follow-up 1) and Day 6 (Follow-up 2) - Part 1: SAD
Description: Absolute baseline values and changes from baseline in pulse rate were summarized by treatment and time post-dose. Baseline was defined as the last pre-dose measurement.
Time Frame: Baseline (pre-dose Day 1), 30 minutes, 2 hours, 6 hour, and 12 hours (post-dose Day 1); 24 hours (End of Treatment), Day 3 (Follow-up 1) and Day 6 (Follow-up 2).
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Part 1: PF-07304814 500 mg 24-hours Continuous Infusion | Part 1: PF-07304814 250 mg 24-hours Continuous Infusion | Part 1: 500 mg Placebo 24-hours Continuous Infusion | Part 1: 250 mg Placebo 24-hours Continuous Infusion
Number analyzed (Participants) | 2 | 2 | 2 | 2
bpm
  Pulse rate: Baseline | 83.0 (2.83) | 74.5 (4.95) | 66.0 (16.97) | 75.5 (6.36)
  Pulse rate: Change from Baseline: Day 1 - 30 minutes: number analyzed (Participants) | 1 | 1 | 1 | 2
  Pulse rate: Change from Baseline: Day 1 - 30 minutes | 1.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 10.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -1.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 6.5 (0.71)
  Pulse rate: Change from Baseline: Day 1 - 2 hours: number analyzed (Participants) | 1 | 2 | 1 | 2
  Pulse rate: Change from Baseline: Day 1 - 2 hours | -2.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 2.5 (3.54) | -5.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 16.0 (24.04)
  Pulse rate: Change from Baseline: Day 1 - 6 hours: number analyzed (Participants) | 1 | 1 | 1 | 0
  Pulse rate: Change from Baseline: Day 1 - 6 hours | -6.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -8.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -7.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. |
  Pulse rate: Change from Baseline: Day 1 - 12 hours: number analyzed (Participants) | 1 | 2 | 2 | 2
  Pulse rate: Change from Baseline: Day 1 - 12 hours | -12.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 0.0 (0.00) | -11.0 (1.41) | 6.0 (7.07)
  Pulse rate: Change from Baseline: End of Treatment: number analyzed (Participants) | 2 | 2 | 2 | 1
  Pulse rate: Change from Baseline: End of Treatment | -5.5 (0.71) | -4.5 (17.68) | 2.5 (10.61) | -17.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  Pulse rate: Change from Baseline: Follow Up 1: number analyzed (Participants) | 2 | 2 | 2 | 1
  Pulse rate: Change from Baseline: Follow Up 1 | -2.5 (7.78) | -7.0 (1.41) | -1.0 (1.41) | 15.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  Pulse rate: Change from Baseline: Follow Up 2: number analyzed (Participants) | 1 | 1 | 1 | 2
  Pulse rate: Change from Baseline: Follow Up 2 | 4.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 3.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 5.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 5.0 (9.90)

10. Primary Outcome: Summary of Baseline and Change From Baseline in Pulse Rate at Day 2, 3, 4, 5, and 6 (120 Hours), Day 7 (Follow-up 1), Day 10 (Follow-up 2), Day 14 (Follow-up 3), Between Day 34-41 (Follow-up 4), and/or Early Termination - Part 2: MAD
Description: as for outcome 9
Time Frame: Baseline (pre-dose Day 1); Day 2, 3, 4, 5; 120 hours (End of Treatment), Day 7 (Follow-up 1), Day 10 (Follow-up 2), Day 14 (Follow-up 3), Follow-up 4 (between Day 34-41) and/or early termination (ET).
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Part 2: PF-07304814 500 mg 120-hours Continuous Infusion | Part 2: PF-07304814 250 mg 120-hours Continuous Infusion | Part 2: Placebo 120-hours Continuous Infusion
Number analyzed (Participants) | 6 | 7 | 4
bpm
  Pulse rate: Baseline | 74.2 (10.59) | 80.9 (13.15) | 90.3 (30.38)
  Pulse rate: Change from Baseline: Day 2 | -4.0 (16.82) | -5.4 (10.64) | -1.5 (4.12)
  Pulse rate: Change from Baseline: Day 3 | 3.5 (11.52) | -6.6 (20.90) | -3.0 (8.60)
  Pulse rate: Change from Baseline: Day 4: number analyzed (Participants) | 6 | 7 | 3
  Pulse rate: Change from Baseline: Day 4 | -6.0 (17.47) | -10.6 (10.39) | -18.3 (24.79)
  Pulse rate: Change from Baseline: Day 5: number analyzed (Participants) | 6 | 7 | 3
  Pulse rate: Change from Baseline: Day 5 | -2.3 (11.11) | -8.4 (12.61) | -12.0 (22.07)
  Pulse rate: Change from Baseline: End of Treatment: number analyzed (Participants) | 6 | 7 | 3
  Pulse rate: Change from Baseline: End of Treatment | -7.8 (20.65) | -9.1 (16.34) | -19.7 (45.39)
  Pulse rate: Change from Baseline: Early Termination: number analyzed (Participants) | 0 | 0 | 1
  Pulse rate: Change from Baseline: Early Termination |  |  | -3.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed
  Pulse rate: Change from Baseline: Follow Up 1 | -1.3 (9.93) | -9.7 (12.58) | -11.3 (32.46)
  Pulse rate: Change from Baseline: Follow Up 2: number analyzed (Participants) | 4 | 1 | 2
  Pulse rate: Change from Baseline: Follow Up 2 | 13.0 (9.83) | -38.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed | -25.5 (24.75)
  Pulse rate: Change from Baseline: Follow Up 3: number analyzed (Participants) | 4 | 2 | 3
  Pulse rate: Change from Baseline: Follow Up 3 | 8.8 (10.24) | 6.0 (29.70) | -7.7 (28.36)
  Pulse rate: Change from Baseline: Follow Up 4: number analyzed (Participants) | 2 | 3 | 1
  Pulse rate: Change from Baseline: Follow Up 4 | 12.0 (12.73) | 8.3 (24.95) | 12.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed

11. Primary Outcome: Summary of Baseline and Change From Baseline in Temperature at Day 1 (30 Minutes, 2 Hours, 6 Hour, and 12 Hours; 24 Hours [End of Treatment]), Day 3 (Follow-up 1) and Day 6 (Follow-up 2) - Part 1: SAD
Description: Absolute baseline values and changes from baseline in temperature were summarized by treatment and time post-dose. Baseline was defined as the last pre-dose measurement.
Time Frame: Baseline (pre-dose Day 1); 30 minutes, 2 hours, 6 hour, and 12 hours (post-dose Day1); 24 hours (End of Treatment), Day 3 (Follow-up 1) and Day 6 (Follow-up 2).
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Part 1: PF-07304814 500 mg 24-hours Continuous Infusion | Part 1: PF-07304814 250 mg 24-hours Continuous Infusion | Part 1: 500 mg Placebo 24-hours Continuous Infusion | Part 1: 250 mg Placebo 24-hours Continuous Infusion
Number analyzed (Participants) | 2 | 2 | 2 | 2
Degree Celsius
  Temperature: Baseline | 37.6 (0.14) | 37.0 (0.28) | 36.5 (0.14) | 37.1 (0.99)
  Temperature: Change from Baseline: Day 1 - 30 minutes | 0.2 (0.21) | -0.2 (0.21) | 0.1 (0.07) | 0.2 (0.00)
  Temperature: Change from Baseline: Day 1 - 2 hours | 0.1 (0.49) | -0.1 (0.07) | 0.1 (0.14) | -0.1 (0.57)
  Temperature: Change from Baseline: Day 1 - 6 hours | -0.4 (0.28) | 0.0 (0.14) | 0.2 (0.07) | 0.1 (0.71)
  Temperature: Change from Baseline: Day 1 - 12 hours | -0.1 (0.99) | -0.5 (0.14) | 0.1 (0.00) | 0.7 (0.42)
  Temperature: Change from Baseline: End of Treatment: number analyzed (Participants) | 2 | 1 | 2 | 2
  Temperature: Change from Baseline: End of Treatment | -0.7 (0.64) | -0.1 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 0.3 (0.35) | 0.3 (0.64)
  Temperature: Change from Baseline: Follow Up 1 | -0.9 (0.78) | -0.7 (0.07) | 0.3 (0.07) | -0.3 (0.85)
  Temperature: Change from Baseline: Follow Up 2: number analyzed (Participants) | 1 | 1 | 1 | 2
  Temperature: Change from Baseline: Follow Up 2 | -0.9 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 2.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 0.3 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 0.1 (0.35)

12. Primary Outcome: Summary of Baseline and Change From Baseline in Temperature at Day 2, 3, 4, 5, and 6 (120 Hours), Day 7 (Follow-up 1), Day 10 (Follow-up 2), Day 14 (Follow-up 3), Between Day 34-41 (Follow-up 4), and/or Early Termination - Part 2: MAD
Description: as for outcome 11
Time Frame: as for outcome 10
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Part 2: PF-07304814 500 mg 120-hours Continuous Infusion | Part 2: PF-07304814 250 mg 120-hours Continuous Infusion | Part 2: Placebo 120-hours Continuous Infusion
Number analyzed (Participants) | 6 | 7 | 4
Degree Celsius
  Temperature: Baseline | 36.7 (0.79) | 36.7 (0.35) | 36.3 (0.73)
  Temperature: Change from Baseline: Day 2 | -0.4 (0.88) | -0.3 (0.50) | 0.2 (0.29)
  Temperature: Change from Baseline: Day 3 | -0.2 (0.84) | -0.3 (0.43) | 0.1 (0.43)
  Temperature: Change from Baseline: Day 4: number analyzed (Participants) | 6 | 7 | 3
  Temperature: Change from Baseline: Day 4 | -0.3 (0.91) | -0.4 (0.45) | 0.0 (0.40)
  Temperature: Change from Baseline: Day 5: number analyzed (Participants) | 6 | 7 | 3
  Temperature: Change from Baseline: Day 5 | -0.4 (0.97) | -0.6 (0.60) | 0.4 (0.55)
  Temperature: Change from Baseline: End of Treatment: number analyzed (Participants) | 6 | 7 | 3
  Temperature: Change from Baseline: End of Treatment | -0.4 (0.91) | -0.6 (0.59) | 0.5 (0.45)
  Temperature: Change from Baseline: Early Termination: number analyzed (Participants) | 0 | 0 | 1
  Temperature: Change from Baseline: Early Termination |  |  | -0.3 (NA) — Standard deviation was not applicable because only 1 participant was analyzed
  Temperature: Change from Baseline: Follow Up 1: number analyzed (Participants) | 6 | 7 | 3
  Temperature: Change from Baseline: Follow Up 1 | -0.4 (0.91) | -0.6 (0.46) | 0.7 (0.17)
  Temperature: Change from Baseline: Follow Up 2: number analyzed (Participants) | 4 | 1 | 2
  Temperature: Change from Baseline: Follow Up 2 | -0.1 (1.21) | -0.1 (NA) — Standard deviation was not applicable because only 1 participant was analyzed | 0.7 (0.57)
  Temperature: Change from Baseline: Follow Up 3: number analyzed (Participants) | 4 | 2 | 3
  Temperature: Change from Baseline: Follow Up 3 | -0.4 (1.05) | -0.1 (0.21) | 0.7 (1.08)
  Temperature: Change from Baseline: Follow Up 4: number analyzed (Participants) | 2 | 3 | 1
  Temperature: Change from Baseline: Follow Up 4 | -1.0 (0.64) | 0.2 (0.67) | -0.2 (NA) — Standard deviation was not applicable because only 1 participant was analyzed

13. Primary Outcome: Summary of Baseline and Change From Baseline in Respiratory Rate at Day 1 (30 Minutes, 2 Hours, 6 Hour, and 12 Hours; 24 Hours [End of Treatment]), Day 3 (Follow-up 1) and Day 6 (Follow-up 2) - Part 1: SAD
Description: Absolute baseline values and changes from baseline in respiratory rate were summarized by treatment and time post-dose. Baseline was defined as the last pre-dose measurement.
Time Frame: as for outcome 11
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Part 1: PF-07304814 500 mg 24-hours Continuous Infusion | Part 1: PF-07304814 250 mg 24-hours Continuous Infusion | Part 1: 500 mg Placebo 24-hours Continuous Infusion | Part 1: 250 mg Placebo 24-hours Continuous Infusion
Number analyzed (Participants) | 2 | 2 | 2 | 2
breaths per minute
  Respiratory rate: Baseline | 21.0 (1.41) | 20.5 (3.54) | 23.0 (7.07) | 20.0 (2.83)
  Respiratory rate: Change from Baseline: Day 1 - 30 minutes: number analyzed (Participants) | 1 | 2 | 2 | 2
  Respiratory rate: Change from Baseline: Day 1 - 30 minutes | 0.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -1.0 (4.24) | -1.0 (1.41) | -0.5 (0.71)
  Respiratory rate: Change from Baseline: Day 1 - 2 hours: number analyzed (Participants) | 1 | 2 | 2 | 2
  Respiratory rate: Change from Baseline: Day 1 - 2 hours | 0.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -1.0 (4.24) | -1.0 (1.41) | 6.5 (7.78)
  Respiratory rate: Change from Baseline: Day 1 - 6 hours: number analyzed (Participants) | 1 | 2 | 2 | 0
  Respiratory rate: Change from Baseline: Day 1 - 6 hours | -2.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -0.5 (0.71) | -0.5 (0.71) |
  Respiratory rate: Change from Baseline: Day 1 - 12 hours | -1.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -5.5 (10.61) | -2.5 (4.95) | 0.0 (0.00)
  Respiratory rate: Change from Baseline: End of Treatment: number analyzed (Participants) | 2 | 2 | 2 | 1
  Respiratory rate: Change from Baseline: End of Treatment | -2.5 (0.71) | -0.5 (2.12) | 2.5 (3.54) | 7.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  Respiratory rate: Change from Baseline: Follow Up 1: number analyzed (Participants) | 2 | 2 | 2 | 1
  Respiratory rate: Change from Baseline: Follow Up 1 | -4.0 (2.83) | 0.5 (7.78) | -3.5 (4.95) | -4.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  Respiratory rate: Change from Baseline: Follow Up 2: number analyzed (Participants) | 1 | 1 | 1 | 2
  Respiratory rate: Change from Baseline: Follow Up 2 | -8.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 4.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -8.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -2.0 (5.66)

14. Primary Outcome: Summary of Baseline and Change From Baseline in Respiratory Rate at Day 2, 3, 4, 5, and 6 (120 Hours), Day 7 (Follow-up 1), Day 10 (Follow-up 2), Day 14 (Follow-up 3), Between Day 34-41 (Follow-up 4), and/or Early Termination - Part 2: MAD
Description: as for outcome 13
Time Frame: as for outcome 10
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 2: PF-07304814 500 mg 120-hours Continuous Infusion | Part 2: PF-07304814 250 mg 120-hours Continuous Infusion | Part 2: Placebo 120-hours Continuous Infusion
Number analyzed (Participants) | 6 | 7 | 4
Breaths per minute
  Respiratory rate: Baseline | 23.5 (3.45) | 22.4 (5.59) | 21.0 (4.69)
  Respiratory rate: Change from Baseline: Day 2 | -3.0 (7.10) | -1.7 (7.45) | -0.5 (5.07)
  Respiratory rate: Change from Baseline: Day 3 | 1.0 (8.99) | -3.1 (4.26) | 1.0 (4.97)
  Respiratory rate: Change from Baseline: Day 4: number analyzed (Participants) | 6 | 7 | 3
  Respiratory rate: Change from Baseline: Day 4 | -1.8 (3.76) | -4.0 (5.69) | 4.0 (5.00)
  Respiratory rate: Change from Baseline: Day 5: number analyzed (Participants) | 6 | 7 | 3
  Respiratory rate: Change from Baseline: Day 5 | -2.2 (5.78) | -2.9 (2.04) | -0.7 (2.08)
  Respiratory rate: Change from Baseline: End of Treatment: number analyzed (Participants) | 6 | 7 | 3
  Respiratory rate: Change from Baseline: End of Treatment | -3.3 (4.27) | -2.3 (5.62) | -2.3 (3.51)
  Respiratory rate: Change from Baseline: Early Termination: number analyzed (Participants) | 0 | 0 | 1
  Respiratory rate: Change from Baseline: Early Termination |  |  | -4.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed
  Respiratory rate: Change from Baseline: Follow Up 1: number analyzed (Participants) | 6 | 7 | 3
  Respiratory rate: Change from Baseline: Follow Up 1 | -3.5 (4.55) | -3.9 (4.88) | -3.0 (1.00)
  Respiratory rate: Change from Baseline: Follow Up 2: number analyzed (Participants) | 4 | 1 | 2
  Respiratory rate: Change from Baseline: Follow Up 2 | -5.8 (6.50) | -2.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed | -1.5 (2.12)
  Respiratory rate: Change from Baseline: Follow Up 3: number analyzed (Participants) | 4 | 1 | 3
  Respiratory rate: Change from Baseline: Follow Up 3 | -6.8 (5.74) | -10.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed | 1.3 (10.12)
  Respiratory rate: Change from Baseline: Follow Up 4: number analyzed (Participants) | 2 | 3 | 1
  Respiratory rate: Change from Baseline: Follow Up 4 | -6.0 (5.66) | 1.3 (4.73) | -3.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed

15. Primary Outcome: Summary of Baseline and Change From Baseline in Pulse Oximetry/SpO2 at 24 Hours (End of Treatment), Day 3 (Follow-up 1) and Day 6 (Follow-up 2) - Part 1: SAD
Description: Percent SpO2 values at baseline and changes from baseline were summarized for participants in 3 categories: (1) participants who received supplemental oxygen throughout, (2) participants who received supplemental oxygen at some point during the study, and (3) participants who never received supplemental oxygen. Baseline of pulse oximetry/SpO2 was defined as the last pre-dose measurement.
  SpO2 = arterial oxygen saturation.
Time Frame: Baseline (pre-dose Day 1); Day1-24 hours (End of Treatment), Day 3 (Follow-up 1) and Day 6 (Follow-up 2)
Population: All participants randomly assigned to study intervention and who take at least 1 dose of study intervention for the Part 1. Participants will be analyzed according to the product they actually received.
  Number of Participants analyzed refers to number of participants evaluable for this OM; Number Analyzed refers to number of participants evaluable at the specific time point.
Measure: Mean (Standard Deviation); unit: percentage of SpO2
Arm/Group | Part 1: PF-07304814 500 mg 24-hours Continuous Infusion | Part 1: PF-07304814 250 mg 24-hours Continuous Infusion | Part 1: 500 mg Placebo 24-hours Continuous Infusion | Part 1: 250 mg Placebo 24-hours Continuous Infusion
Number analyzed (Participants) | 2 | 2 | 2 | 2
percentage of SpO2
  Baseline: Oxygen Received Throughout: number analyzed (Participants) | 1 | 1 | 1 | 2
  Baseline: Oxygen Received Throughout | 92.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 90.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 98.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 94.5 (0.71)
  Baseline: Oxygen Received at Some Point During Study: number analyzed (Participants) | 0 | 1 | 1 | 0
  Baseline: Oxygen Received at Some Point During Study |  | 91.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 95.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. |
  Baseline: Oxygen Never Received: number analyzed (Participants) | 1 | 0 | 0 | 0
  Baseline: Oxygen Never Received | 93.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. |  |  |
  Change from Baseline: End of Treatment: Oxygen Received Throughout:: number analyzed (Participants) | 1 | 1 | 1 | 2
  Change from Baseline: End of Treatment: Oxygen Received Throughout: | 3.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 5.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 0.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -0.5 (0.71)
  Change from Baseline: End of Treatment: Oxygen Received at Some Point During Study: number analyzed (Participants) | 0 | 1 | 1 | 0
  Change from Baseline: End of Treatment: Oxygen Received at Some Point During Study |  | 5.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -4.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. |
  Change from Baseline: End of Treatment: Oxygen Never Received: number analyzed (Participants) | 1 | 0 | 0 | 0
  Change from Baseline: End of Treatment: Oxygen Never Received | 1.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. |  |  |
  Change from Baseline: Follow Up 1: Oxygen Received Throughout: number analyzed (Participants) | 1 | 1 | 1 | 1
  Change from Baseline: Follow Up 1: Oxygen Received Throughout | 3.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 1.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 0.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 0.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  Change from Baseline: Follow Up 1: Oxygen Received at Some Point During Study: number analyzed (Participants) | 0 | 1 | 1 | 0
  Change from Baseline: Follow Up 1: Oxygen Received at Some Point During Study |  | 5.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 1.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. |
  Change from Baseline: Follow Up 1: Oxygen Never Received: number analyzed (Participants) | 1 | 0 | 0 | 0
  Change from Baseline: Follow Up 1: Oxygen Never Received | 1.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. |  |  |
  Change from Baseline: Follow Up 2: Oxygen Received Throughout: number analyzed (Participants) | 1 | 1 | 1 | 2
  Change from Baseline: Follow Up 2: Oxygen Received Throughout | 0.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 5.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -5.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -1.5 (0.71)
  Change from Baseline: Follow Up 2: Oxygen Received at Some Point During Study: number analyzed (Participants) | 0 | 0 | 0 | 0
  Change from Baseline: Follow Up 2: Oxygen Never Received: number analyzed (Participants) | 0 | 0 | 0 | 0

16. Primary Outcome: Summary of Baseline and Change From Baseline in Pulse Oximetry/SpO2 at Day 2, 3, 4, 5; 6 (120hours), Day 7 (Follow-up 1), Day 10 (Follow-up 2), Day 14 (Follow-up 3), Follow-up 4 (Between Day 34-41), and/or Early Termination-Part 2: MAD
Description: as for outcome 15
Time Frame: Baseline (pre-dose Day 1); Day 2, 3, 4, 5; 120 hours (End of Treatment), Day 7 (Follow-up 1), Day 10 (Follow-up 2), Day 14 (Follow-up 3), Follow-up 4 (between Day 34-41), and/or early termination (ET).
Population: All participants randomly assigned to study intervention and who take at least 1 dose of study intervention for the Part 2. Participants will be analyzed according to the product they actually received.
  Number of Participants analyzed refers to number of participants evaluable for this OM; Number Analyzed refers to number of participants evaluable at the specific time point.
Measure: Mean (Standard Deviation); unit: percentage of SpO2
Arm/Group | Part 2: PF-07304814 500 mg 120-hours Continuous Infusion | Part 2: PF-07304814 250 mg 120-hours Continuous Infusion | Part 2: Placebo 120-hours Continuous Infusion
Number analyzed (Participants) | 6 | 7 | 4
percentage of SpO2
  Baseline: Oxygen Received Throughout: number analyzed (Participants) | 4 | 3 | 1
  Baseline: Oxygen Received Throughout | 93.3 (3.77) | 96.3 (0.58) | 60.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  Baseline: Oxygen Received at Some Point During Study: number analyzed (Participants) | 2 | 3 | 3
  Baseline: Oxygen Received at Some Point During Study | 97.0 (0.00) | 96.0 (2.65) | 97.3 (0.58)
  Baseline: Oxygen Never Received: number analyzed (Participants) | 0 | 1 | 0
  Baseline: Oxygen Never Received |  | 98.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. |
  Change from Baseline: Day 2: Oxygen Received Throughout: number analyzed (Participants) | 4 | 3 | 1
  Change from Baseline: Day 2: Oxygen Received Throughout | 2.0 (3.74) | -3.3 (2.08) | 34.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  Change from Baseline: Day 2: Oxygen Received at Some Point During Study: number analyzed (Participants) | 2 | 3 | 3
  Change from Baseline: Day 2: Oxygen Received at Some Point During Study | 1.0 (0.00) | -1.0 (1.0) | -2.7 (2.08)
  Change from Baseline: Day 2: Oxygen Never Received: number analyzed (Participants) | 0 | 1 | 0
  Change from Baseline: Day 2: Oxygen Never Received |  | 2.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. |
  Change from Baseline: Day 3: Oxygen Received Throughout: number analyzed (Participants) | 4 | 3 | 1
  Change from Baseline: Day 3: Oxygen Received Throughout | 1.3 (3.77) | -2.3 (2.08) | 31.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  Change from Baseline: Day 3: Oxygen Received at Some Point During Study: number analyzed (Participants) | 2 | 3 | 3
  Change from Baseline: Day 3: Oxygen Received at Some Point During Study | -2.0 (2.83) | 0.0 (1.00) | -1.0 (1.0)
  Change from Baseline: Day 3: Oxygen Never Received: number analyzed (Participants) | 0 | 1 | 0
  Change from Baseline: Day 3: Oxygen Never Received |  | -3.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. |
  Change from Baseline: Day 4: Oxygen Received Throughout: number analyzed (Participants) | 4 | 3 | 1
  Change from Baseline: Day 4: Oxygen Received Throughout | 2.0 (2.45) | -0.7 (2.52) | 29.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  Change from Baseline: Day 4: Oxygen Received at Some Point During Study: number analyzed (Participants) | 2 | 3 | 2
  Change from Baseline: Day 4: Oxygen Received at Some Point During Study | -1.0 (0.00) | -0.7 (0.58) | -3.5 (2.12)
  Change from Baseline: Day 4: Oxygen Never Received: number analyzed (Participants) | 0 | 1 | 0
  Change from Baseline: Day 4: Oxygen Never Received |  | -3.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. |
  Change from Baseline: Day 5: Oxygen Received Throughout: number analyzed (Participants) | 4 | 3 | 1
  Change from Baseline: Day 5: Oxygen Received Throughout | 3.0 (4.08) | -1.3 (3.79) | 25.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  Change from Baseline: Day 5: Oxygen Received at Some Point During Study: number analyzed (Participants) | 2 | 3 | 2
  Change from Baseline: Day 5: Oxygen Received at Some Point During Study | -1.5 (0.71) | -1.3 (2.08) | -5.5 (3.54)
  Change from Baseline: Day 5: Oxygen Never Received: number analyzed (Participants) | 0 | 1 | 0
  Change from Baseline: Day 5: Oxygen Never Received |  | -2.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. |
  Change from Baseline: End of Treatment: Oxygen Received Throughout: number analyzed (Participants) | 4 | 3 | 1
  Change from Baseline: End of Treatment: Oxygen Received Throughout | 0.8 (3.86) | -1.0 (1.73) | 34.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  Change from Baseline: End of Treatment: Oxygen Received at Some Point During Study: number analyzed (Participants) | 2 | 3 | 2
  Change from Baseline: End of Treatment: Oxygen Received at Some Point During Study | 0.0 (2.83) | 0.3 (2.08) | -5.5 (0.71)
  Change from Baseline: End of Treatment: Oxygen Never Received: number analyzed (Participants) | 0 | 1 | 0
  Change from Baseline: End of Treatment: Oxygen Never Received |  | 0.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. |
  Change from Baseline: Early Termination: Oxygen Received Throughout: number analyzed (Participants) | 0 | 0 | 0
  Change from Baseline: Early Termination: Oxygen Received at Some Point During Study: number analyzed (Participants) | 0 | 0 | 1
  Change from Baseline: Early Termination: Oxygen Received at Some Point During Study |  |  | -1.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  Change from Baseline: Early Termination: Oxygen Never Received: number analyzed (Participants) | 0 | 0 | 0
  Change from Baseline: Follow Up 1: Oxygen Received Throughout: number analyzed (Participants) | 4 | 3 | 1
  Change from Baseline: Follow Up 1: Oxygen Received Throughout | 2.0 (2.45) | -1.0 (0.00) | 36.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  Change from Baseline: Follow Up 1: Oxygen Received at Some Point During Study: number analyzed (Participants) | 2 | 3 | 2
  Change from Baseline: Follow Up 1: Oxygen Received at Some Point During Study | -2.5 (0.71) | 0.0 (1.73) | -3.0 (2.83)
  Change from Baseline: Follow Up 1: Oxygen Never Received: number analyzed (Participants) | 0 | 1 | 0
  Change from Baseline: Follow Up 1: Oxygen Never Received |  | -1.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. |
  Change from Baseline: Follow Up 2: Oxygen Received Throughout: number analyzed (Participants) | 3 | 1 | 1
  Change from Baseline: Follow Up 2: Oxygen Received Throughout | 3.3 (4.04) | -2.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 31.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  Change from Baseline: Follow Up 2: Oxygen Received at Some Point During Study: number analyzed (Participants) | 1 | 0 | 1
  Change from Baseline: Follow Up 2: Oxygen Received at Some Point During Study | -2.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. |  | 1.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  Change from Baseline: Follow Up 2: Oxygen Never Received: number analyzed (Participants) | 0 | 0 | 0
  Change from Baseline: Follow Up 3: Oxygen Received Throughout: number analyzed (Participants) | 3 | 1 | 1
  Change from Baseline: Follow Up 3: Oxygen Received Throughout | 3.7 (4.04) | -2.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 31.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  Change from Baseline: Follow Up 3: Oxygen Received at Some Point During Study: number analyzed (Participants) | 1 | 1 | 2
  Change from Baseline: Follow Up 3: Oxygen Received at Some Point During Study | 0.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 2.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 0.5 (0.71)
  Change from Baseline: Follow Up 3: Oxygen Never Received: number analyzed (Participants) | 0 | 0 | 0
  Change from Baseline: Follow Up 4: Oxygen Received Throughout: number analyzed (Participants) | 2 | 2 | 0
  Change from Baseline: Follow Up 4: Oxygen Received Throughout | 3.0 (1.41) | -0.5 (3.54) |
  Change from Baseline: Follow Up 4: Oxygen Received at Some Point During Study: number analyzed (Participants) | 0 | 1 | 1
  Change from Baseline: Follow Up 4: Oxygen Received at Some Point During Study |  | 1.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -3.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  Change from Baseline: Follow Up 4: Oxygen Never Received: number analyzed (Participants) | 0 | 0 | 0

17. Primary Outcome: Summary of Baseline and Change From Baseline in ECG Mean Heart Rate at Day 1 (30 Minutes, 2 Hours, 6 Hour, and 12 Hours; 24 Hours [End of Treatment]), Day 3 (Follow-up 1) and Day 6 (Follow-up 2) - Part 1: SAD
Description: The average of the triplicate readings collected at each assessment time was calculated for each ECG parameter. Baseline was defined as the average (if possible) of the triplicate pre-dose recordings on Day 1. Only centrally read ECG data was used.
Time Frame: as for outcome 11
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention for Part 1. Participants were analyzed according to the product they received.
  Number of Participants analyzed refers to number of participants evaluable for this OM; Number Analyzed refers to number of participants evaluable at the specific time point.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1: PF-07304814 500 mg 24-hours Continuous Infusion | Part 1: PF-07304814 250 mg 24-hours Continuous Infusion | Part 1: 500 mg Placebo 24-hours Continuous Infusion | Part 1: 250 mg Placebo 24-hours Continuous Infusion
Number analyzed (Participants) | 2 | 2 | 2 | 2
Beats per minute
  ECG mean heart rate: Baseline | 87.5 (3.54) | 71.5 (4.95) | 66.0 (15.56) | 71.0 (7.07)
  ECG mean heart rate: Change from Baseline: Day 1 - 30 minutes: number analyzed (Participants) | 2 | 0 | 2 | 0
  ECG mean heart rate: Change from Baseline: Day 1 - 30 minutes | -3.5 (3.54) |  | -5.5 (0.71) |
  ECG mean heart rate: Change from Baseline: Day 1 - 2 hours: number analyzed (Participants) | 2 | 0 | 2 | 0
  ECG mean heart rate: Change from Baseline: Day 1 - 2 hours | 2.0 (8.49) |  | -4.0 (2.83) |
  ECG mean heart rate: Change from Baseline: Day 1 - 6 hours | -12.5 (4.95) | 2.5 (0.71) | -13.5 (9.19) | 7.5 (13.44)
  ECG mean heart rate: Change from Baseline: Day 1 - 12 hours | -7.0 (11.31) | 3.0 (5.66) | -9.5 (3.54) | 8.5 (10.61)
  ECG mean heart rate: Change from Baseline: End of Treatment | -7.0 (5.66) | -9.0 (7.07) | 2.5 (10.61) | -4.0 (2.83)
  ECG mean heart rate: Change from Baseline: Follow Up 1: number analyzed (Participants) | 2 | 1 | 2 | 2
  ECG mean heart rate: Change from Baseline: Follow Up 1 | -8.0 (11.31) | -2.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -3.5 (0.71) | 8.0 (5.66)
  ECG mean heart rate: Change from Baseline: Follow Up 2: number analyzed (Participants) | 1 | 1 | 1 | 1
  ECG mean heart rate: Change from Baseline: Follow Up 2 | -14.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 1.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 1.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -8.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.

18. Primary Outcome: Summary of Baseline and Change From Baseline in ECG Mean Heart Rate at Day 2, 3, 5, 6 (120 Hours), Day 7 (Follow-up 1), Day 10 (Follow-up 2), Day 14 (Follow-up 3), Follow-up 4 (Between Day 34-41) and/or Early Termination- Part 2: MAD
Description: as for outcome 17
Time Frame: Baseline (pre-dose Day 1); Day 2, 3, 5; 120 hours (End of Treatment), Day 7 (Follow-up 1), Day 10 (Follow-up 2), Day 14 (Follow-up 3), Follow-up 4 (between Day 34-41), and/or early termination(ET)
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention for Part 2. Participants were analyzed according to the product they received.
  Number of Participants analyzed refers to number of participants evaluable for this OM; Number Analyzed refers to number of participants evaluable at the specific time point.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2: PF-07304814 500 mg 120-hours Continuous Infusion | Part 2: PF-07304814 250 mg 120-hours Continuous Infusion | Part 2: Placebo 120-hours Continuous Infusion
Number analyzed (Participants) | 6 | 7 | 4
Beats per minute
  ECG mean heart rate: Baseline | 70.2 (9.02) | 80.1 (11.29) | 85.0 (41.16)
  ECG mean heart rate: Change from Baseline: Day 2: number analyzed (Participants) | 6 | 6 | 3
  ECG mean heart rate: Change from Baseline: Day 2 | -4.7 (8.52) | -6.0 (18.90) | -0.7 (2.08)
  ECG mean heart rate: Change from Baseline: Day 3: number analyzed (Participants) | 6 | 6 | 4
  ECG mean heart rate: Change from Baseline: Day 3 | -8.7 (15.49) | -12.0 (15.01) | -7.5 (18.91)
  ECG mean heart rate: Change from Baseline: Day 5: number analyzed (Participants) | 6 | 7 | 3
  ECG mean heart rate: Change from Baseline: Day 5 | -6.7 (13.28) | -9.0 (8.04) | -13.7 (27.61)
  ECG mean heart rate: Change from Baseline: End of Treatment: number analyzed (Participants) | 6 | 7 | 3
  ECG mean heart rate: Change from Baseline: End of Treatment | -8.7 (16.65) | -8.4 (13.46) | -15.0 (42.79)
  ECG mean heart rate: Change from Baseline: Early Termination: number analyzed (Participants) | 0 | 0 | 1
  ECG mean heart rate: Change from Baseline: Early Termination |  |  | 9.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  ECG mean heart rate: Change from Baseline: Follow Up 1: number analyzed (Participants) | 5 | 7 | 3
  ECG mean heart rate: Change from Baseline: Follow Up 1 | 2.8 (17.73) | -6.9 (8.63) | 21.0 (10.44)
  ECG mean heart rate: Change from Baseline: Follow Up 2: number analyzed (Participants) | 4 | 1 | 1
  ECG mean heart rate: Change from Baseline: Follow Up 2 | 7.0 (12.68) | -26.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 2.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  ECG mean heart rate: Change from Baseline: Follow Up 3: number analyzed (Participants) | 4 | 2 | 1
  ECG mean heart rate: Change from Baseline: Follow Up 3 | 8.5 (12.07) | -12.5 (16.26) | 6.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  ECG mean heart rate: Change from Baseline: Follow Up 4: number analyzed (Participants) | 1 | 3 | 1
  ECG mean heart rate: Change from Baseline: Follow Up 4 | -6.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 8.0 (21.38) | 21.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.

19. Primary Outcome: Summary of Baseline and Change From Baseline in PR, QRS, QT and QTcF Intervals at Day 1 (30 Minutes, 2 Hours, 6 Hour, and 12 Hours; 24 Hours [End of Treatment]), Day 3 (Follow-up 1) and Day 6 (Follow-up 2) - Part 1: SAD
Description: as for outcome 17
Time Frame: as for outcome 11
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Millisecond
Arm/Group | Part 1: PF-07304814 500 mg 24-hours Continuous Infusion | Part 1: PF-07304814 250 mg 24-hours Continuous Infusion | Part 1: 500 mg Placebo 24-hours Continuous Infusion | Part 1: 250 mg Placebo 24-hours Continuous Infusion
Number analyzed (Participants) | 2 | 2 | 2 | 2
Millisecond
  PR interval: Baseline | 153.0 (5.66) | 165.0 (29.70) | 171.0 (16.97) | 183.5 (10.61)
  PR interval: Change from Baseline: Day 1 - 30 minutes: number analyzed (Participants) | 2 | 0 | 2 | 0
  PR interval: Change from Baseline: Day 1 - 30 minutes | -7.0 (1.41) |  | -1.5 (0.71) |
  PR interval: Change from Baseline: Day 1 - 2 hours: number analyzed (Participants) | 2 | 0 | 2 | 0
  PR interval: Change from Baseline: Day 1 - 2 hours | -6.0 (14.14) |  | -2.5 (2.12) |
  PR interval: Change from Baseline: Day 1 - 6 hours | -3.5 (4.95) | -1.5 (7.78) | -2.5 (4.95) | -14.5 (4.95)
  PR interval: Change from Baseline: Day 1 - 12 hours | -4.0 (11.31) | -11.0 (19.80) | 0.5 (3.54) | -19.5 (4.95)
  PR interval: Change from Baseline: End of Treatment | -8.0 (2.83) | 1.5 (10.61) | -7.5 (6.36) | -7.0 (5.66)
  PR interval: Change from Baseline: Follow Up 1: number analyzed (Participants) | 2 | 1 | 2 | 2
  PR interval: Change from Baseline: Follow Up 1 | -3.5 (12.02) | 5.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -2.0 (12.73) | -16.5 (6.36)
  PR interval: Change from Baseline: Follow Up 2: number analyzed (Participants) | 1 | 1 | 1 | 1
  PR interval: Change from Baseline: Follow Up 2 | 9.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -1.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -7.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -11.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  QRS interval: Baseline | 92.5 (2.12) | 99.0 (4.24) | 95.0 (8.49) | 103.0 (4.24)
  QRS interval: Change from Baseline: Day 1 - 30 minutes: number analyzed (Participants) | 2 | 0 | 2 | 0
  QRS interval: Change from Baseline: Day 1 - 30 minutes | -2.0 (5.66) |  | 1.0 (2.83) |
  QRS interval: Change from Baseline: Day 1 - 2 hours: number analyzed (Participants) | 2 | 0 | 2 | 0
  QRS interval: Change from Baseline: Day 1 - 2 hours | -2.5 (0.71) |  | 1.0 (1.41) |
  QRS interval: Change from Baseline: Day 1 - 6 hours | -2.5 (2.12) | -3.0 (12.73) | -2.0 (2.83) | 0.0 (1.41)
  QRS interval: Change from Baseline: Day 1 - 12 hours | -2.5 (0.71) | 0.0 (5.66) | -3.0 (0.00) | -0.5 (3.54)
  QRS interval: Change from Baseline: End of Treatment | 1.5 (6.36) | 0.0 (1.41) | 0.0 (4.24) | 0.5 (0.71)
  QRS interval: Change from Baseline: Follow Up 1: number analyzed (Participants) | 2 | 1 | 2 | 2
  QRS interval: Change from Baseline: Follow Up 1 | 1.0 (0.00) | -1.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -5.0 (1.41) | 0.0 (2.83)
  QRS interval: Change from Baseline: Follow Up 2: number analyzed (Participants) | 1 | 1 | 1 | 1
  QRS interval: Change from Baseline: Follow Up 2 | -1.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -2.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 2.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 1.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  QT interval: Baseline | 348.5 (30.41) | 401.0 (48.08) | 397.5 (30.41) | 389.0 (22.63)
  QT interval: Change from Baseline: Day 1 - 30 minutes: number analyzed (Participants) | 2 | 0 | 2 | 0
  QT interval: Change from Baseline: Day 1 - 30 minutes | 5.5 (21.92) |  | 1.0 (12.73) |
  QT interval: Change from Baseline: Day 1 - 2 hours: number analyzed (Participants) | 2 | 0 | 2 | 0
  QT interval: Change from Baseline: Day 1 - 2 hours | -3.5 (12.02) |  | -1.0 (14.14) |
  QT interval: Change from Baseline: Day 1 - 6 hours | 24.5 (10.61) | -16.5 (24.75) | 19.5 (38.89) | -13.5 (28.99)
  QT interval: Change from Baseline: Day 1 - 12 hours | 28.5 (30.41) | -1.0 (1.41) | 30.0 (19.80) | -20.0 (28.28)
  QT interval: Change from Baseline: End of Treatment | 28.0 (16.97) | 28.5 (36.06) | -6.5 (37.48) | 15.0 (11.31)
  QT interval: Change from Baseline: Follow Up 1: number analyzed (Participants) | 2 | 1 | 2 | 2
  QT interval: Change from Baseline: Follow Up 1 | 28.5 (26.16) | 2.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -12.0 (15.56) | -8.5 (2.12)
  QT interval: Change from Baseline: Follow Up 2: number analyzed (Participants) | 1 | 1 | 1 | 1
  QT interval: Change from Baseline: Follow Up 2 | 38.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -13.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -23.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 38.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  QTcF: Baseline | 395.0 (28.28) | 423.0 (41.01) | 408.0 (1.41) | 411.5 (10.61)
  QTcF: Change from Baseline: Day 1 - 30 minutes: number analyzed (Participants) | 2 | 0 | 2 | 0
  QTcF: Change from Baseline: Day 1 - 30 minutes | -1.0 (19.80) |  | -10.0 (14.14) |
  QTcF: Change from Baseline: Day 1 - 2 hours: number analyzed (Participants) | 2 | 0 | 2 | 0
  QTcF: Change from Baseline: Day 1 - 2 hours | -2.0 (2.83) |  | -8.5 (9.19) |
  QTcF: Change from Baseline: Day 1 - 6 hours | 7.0 (16.97) | -10.5 (23.33) | -9.5 (21.92) | -1.0 (7.07)
  QTcF: Change from Baseline: Day 1 - 12 hours | 17.5 (12.02) | 5.0 (7.07) | 9.5 (17.68) | -6.0 (9.90)
  QTcF: Change from Baseline: End of Treatment | 18.5 (7.78) | 9.0 (14.14) | 0.5 (16.26) | 6.5 (6.36)
  QTcF: Change from Baseline: Follow Up 1: number analyzed (Participants) | 2 | 1 | 2 | 2
  QTcF: Change from Baseline: Follow Up 1 | 16.0 (8.49) | 1.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -19.0 (15.56) | 6.0 (9.90)
  QTcF: Change from Baseline: Follow Up 2: number analyzed (Participants) | 1 | 1 | 1 | 1
  QTcF: Change from Baseline: Follow Up 2 | 18.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -12.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -21.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 24.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.

20. Primary Outcome: Summary of Baseline and Change From Baseline in PR, QRS, QT and QTcF Intervals at Day 2, 3, 5, 6 (120 Hours), Day 7 (Follow-up 1), Day 10 (Follow-up 2), Day 14 (Follow-up 3), Follow-up 4 (Between Day 34-41) and/or Early Termination- Part 2: MAD
Description: as for outcome 17
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Millisecond
Arm/Group | Part 2: PF-07304814 500 mg 120-hours Continuous Infusion | Part 2: PF-07304814 250 mg 120-hours Continuous Infusion | Part 2: Placebo 120-hours Continuous Infusion
Number analyzed (Participants) | 6 | 7 | 4
Millisecond
  PR interval: Baseline | 145.7 (12.86) | 139.7 (19.14) | 156.0 (28.31)
  PR interval: Change from Baseline: Day 2: number analyzed (Participants) | 6 | 6 | 3
  PR interval: Change from Baseline: Day 2 | 3.8 (14.76) | -5.0 (15.17) | 1.3 (4.51)
  PR interval: Change from Baseline: Day 3: number analyzed (Participants) | 6 | 6 | 3
  PR interval: Change from Baseline: Day 3 | 1.2 (17.88) | -3.2 (9.91) | 6.0 (11.36)
  PR interval: Change from Baseline: Day 5: number analyzed (Participants) | 6 | 7 | 2
  PR interval: Change from Baseline: Day 5 | 5.7 (19.81) | -1.6 (13.50) | -3.0 (14.14)
  PR interval: Change from Baseline: End of Treatment: number analyzed (Participants) | 6 | 7 | 3
  PR interval: Change from Baseline: End of Treatment | 9.3 (15.46) | -0.6 (15.82) | -0.3 (7.64)
  PR interval: Change from Baseline: Early Termination: number analyzed (Participants) | 0 | 0 | 1
  PR interval: Change from Baseline: Early Termination |  |  | -1.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  PR interval: Change from Baseline: Follow Up 1: number analyzed (Participants) | 5 | 7 | 3
  PR interval: Change from Baseline: Follow Up 1 | 7.2 (18.63) | 1.4 (17.86) | -8.0 (18.36)
  PR interval: Change from Baseline: Follow Up 2: number analyzed (Participants) | 4 | 1 | 1
  PR interval: Change from Baseline: Follow Up 2 | 6.8 (28.85) | -30.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -6.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  PR interval: Change from Baseline: Follow Up 3: number analyzed (Participants) | 4 | 2 | 1
  PR interval: Change from Baseline: Follow Up 3 | 12.0 (24.45) | -21.0 (31.11) | -18.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  PR interval: Change from Baseline: Follow Up 4: number analyzed (Participants) | 1 | 3 | 1
  PR interval: Change from Baseline: Follow Up 4 | 15.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -4.0 (19.31) | -23.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  QRS interval: Baseline | 93.7 (4.68) | 93.6 (10.63) | 90.5 (4.43)
  QRS interval: Change from Baseline: Day 2: number analyzed (Participants) | 6 | 6 | 3
  QRS interval: Change from Baseline: Day 2 | 6.7 (7.94) | 1.7 (5.09) | 4.7 (7.09)
  QRS interval: Change from Baseline: Day 3: number analyzed (Participants) | 6 | 6 | 4
  QRS interval: Change from Baseline: Day 3 | -0.7 (3.08) | 3.5 (5.32) | 3.3 (3.30)
  QRS interval: Change from Baseline: Day 5: number analyzed (Participants) | 6 | 7 | 3
  QRS interval: Change from Baseline: Day 5 | 0.7 (2.88) | 3.0 (3.92) | 7.0 (5.29)
  QRS interval: Change from Baseline: End of Treatment: number analyzed (Participants) | 6 | 7 | 3
  QRS interval: Change from Baseline: End of Treatment | 0.3 (3.78) | 5.6 (5.56) | 2.3 (3.51)
  QRS interval: Change from Baseline: Early Termination: number analyzed (Participants) | 0 | 0 | 1
  QRS interval: Change from Baseline: Early Termination |  |  | -3.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  QRS interval: Change from Baseline: Follow Up 1: number analyzed (Participants) | 5 | 7 | 3
  QRS interval: Change from Baseline: Follow Up 1 | 1.0 (4.18) | 4.0 (6.43) | 2.3 (6.35)
  QRS interval: Change from Baseline: Follow Up 2: number analyzed (Participants) | 4 | 1 | 1
  QRS interval: Change from Baseline: Follow Up 2 | 2.3 (4.50) | 16.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 8.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  QRS interval: Change from Baseline: Follow Up 3: number analyzed (Participants) | 4 | 2 | 1
  QRS interval: Change from Baseline: Follow Up 3 | -0.3 (4.86) | 6.0 (5.66) | 15.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  QRS interval: Change from Baseline: Follow Up 4: number analyzed (Participants) | 1 | 3 | 1
  QRS interval: Change from Baseline: Follow Up 4 | -12.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 7.0 (3.61) | 5.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  QT interval: Baseline | 385.5 (24.74) | 366.1 (22.17) | 373.8 (59.57)
  QT interval: Change from Baseline: Day 2: number analyzed (Participants) | 6 | 6 | 3
  QT interval: Change from Baseline: Day 2 | 25.3 (35.59) | 16.2 (48.16) | 8.3 (9.07)
  QT interval: Change from Baseline: Day 3: number analyzed (Participants) | 6 | 6 | 4
  QT interval: Change from Baseline: Day 3 | 27.5 (59.06) | 27.3 (43.01) | 10.0 (37.34)
  QT interval: Change from Baseline: Day 5: number analyzed (Participants) | 6 | 7 | 3
  QT interval: Change from Baseline: Day 5 | 12.5 (31.04) | 29.0 (21.57) | 28.0 (61.54)
  QT interval: Change from Baseline: End of Treatment: number analyzed (Participants) | 6 | 7 | 3
  QT interval: Change from Baseline: End of Treatment | 21.8 (46.10) | 23.3 (31.07) | 8.0 (60.61)
  QT interval: Change from Baseline: Early Termination: number analyzed (Participants) | 0 | 0 | 1
  QT interval: Change from Baseline: Early Termination |  |  | -17.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  QT interval: Change from Baseline: Follow Up 1: number analyzed (Participants) | 5 | 7 | 3
  QT interval: Change from Baseline: Follow Up 1 | -10.2 (39.09) | 20.9 (16.82) | -49.7 (32.59)
  QT interval: Change from Baseline: Follow Up 2: number analyzed (Participants) | 4 | 1 | 1
  QT interval: Change from Baseline: Follow Up 2 | -19.3 (27.00) | 63.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 0.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  QT interval: Change from Baseline: Follow Up 3: number analyzed (Participants) | 4 | 2 | 1
  QT interval: Change from Baseline: Follow Up 3 | -22.0 (22.17) | 24.5 (13.44) | -21.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  QT interval: Change from Baseline: Follow Up 4: number analyzed (Participants) | 1 | 3 | 1
  QT interval: Change from Baseline: Follow Up 4 | 5.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | -4.0 (39.36) | -36.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  QTcF: Baseline | 404.7 (18.13) | 401.3 (10.44) | 405.3 (18.84)
  QTcF: Change from Baseline: Day 2: number analyzed (Participants) | 6 | 6 | 3
  QTcF: Change from Baseline: Day 2 | 17.5 (20.96) | 6.8 (19.75) | 9.0 (7.94)
  QTcF: Change from Baseline: Day 3: number analyzed (Participants) | 6 | 6 | 4
  QTcF: Change from Baseline: Day 3 | 8.3 (27.66) | 8.0 (21.80) | 7.5 (24.19)
  QTcF: Change from Baseline: Day 5: number analyzed (Participants) | 6 | 7 | 3
  QTcF: Change from Baseline: Day 5 | -0.2 (11.82) | 16.4 (20.74) | 19.7 (39.37)
  QTcF: Change from Baseline: End of Treatment: number analyzed (Participants) | 6 | 7 | 3
  QTcF: Change from Baseline: End of Treatment | 3.7 (16.50) | 10.7 (17.93) | -1.3 (15.50)
  QTcF: Change from Baseline: Early Termination: number analyzed (Participants) | 0 | 0 | 1
  QTcF: Change from Baseline: Early Termination |  |  | -1.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  QTcF: Change from Baseline: Follow Up 1: number analyzed (Participants) | 5 | 7 | 3
  QTcF: Change from Baseline: Follow Up 1 | -7.2 (9.09) | 9.1 (18.43) | -15.7 (23.01)
  QTcF: Change from Baseline: Follow Up 2: number analyzed (Participants) | 4 | 1 | 1
  QTcF: Change from Baseline: Follow Up 2 | -5.8 (9.00) | 18.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 9.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  QTcF: Change from Baseline: Follow Up 3: number analyzed (Participants) | 4 | 2 | 1
  QTcF: Change from Baseline: Follow Up 3 | -7.3 (9.54) | 4.5 (13.44) | -7.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.
  QTcF: Change from Baseline: Follow Up 4: number analyzed (Participants) | 1 | 3 | 1
  QTcF: Change from Baseline: Follow Up 4 | -6.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 2.3 (19.43) | 7.0 (NA) — Standard deviation was not applicable because only 1 participant was analyzed.

21. Secondary Outcome: PF-07304814 (Prodrug) and PF-00835231 (Active Moiety) Plasma PK Parameters: Concentration at 24 Hours (End of Infusion) - Part 1: SAD
Description: C24 was defined as concentration at 24 hours. 24-hour PK draw was approximately 4 hours post end of infusion which corresponded to 28 hours.
Time Frame: Pre-dose and 6 hours post-dose on Day 1; 24 hours; 48 hours; and/or early termination.
Population: All participants randomly assigned to study intervention and who take at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest are reported for Part 1: SAD.
  Number of Participants analyzed refers to number of participants evaluable for this OM; Number Analyzed refers to number of participants evaluable at different parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: PF-07304814 500 mg 24-hours Continuous Infusion | Part 1: PF-07304814 250 mg 24-hours Continuous Infusion
Number analyzed (Participants) | 1 | 2
ng/mL
  C24 of PF-07304814 | NA (NA) — Geometric mean and CV is not applicable with n=1. | NA (NA) — Geometric mean and CV is not applicable due to n<3.
  C24 of PF-00835231 | NA (NA) — Geometric mean and CV is not applicable with n=1. | NA (NA) — Geometric mean and CV is not applicable due to n<3.

22. Secondary Outcome: PF-07304814 (Prodrug) and PF-00835231 (Active Moiety) Plasma PK Parameter: Concentration at 120 Hours (End of Infusion) - Part 2: MAD
Description: C120 was defined as concentration at 120 hours. Blood sample collection at approximately at 2 and 6 hours post the end of the infusion, which correspond to approximately 122 hours and 126 hours post the start of infusion.
Time Frame: Pre-dose on Day1; Day 2, 3, 5 and 6 (end of treatment day), 7 (Follow-up 1), and/or early termination.
Population: All participants randomly assigned to study intervention and who take at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest are reported for Part 2: MAD.
  Number of Participants analyzed refers to number of participants evaluable for this OM; Number Analyzed refers to number of participants evaluable at different parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: PF-07304814 500 mg 120-hours Continuous Infusion | Part 2: PF-07304814 250 mg 120-hours Continuous Infusion
Number analyzed (Participants) | 6 | 7
ng/mL
  C120 of PF-07304814: number analyzed (Participants) | 5 | 7
  C120 of PF-07304814 | 197.2 (72) | 91.64 (51)
  C120 of PF-00835231 | 1338 (84) | 800.8 (19)

23. Secondary Outcome: PF-07304814 (Prodrug) and PF-00835231 (Active Moiety) Plasma PK Parameters: Maximum Observed Concentration (Cmax) - Part 2: MAD
Description: Cmax was defined as maximum observed concentration. Blood sample collection at approximately 2 and 6 hours post the end of the infusion, which correspond to approximately 122 hours and 126 hours post the start of infusion.
Time Frame: Pre-dose on Day1; Day 2, 3, 5 and 6 (end of treatment day), 7 (Follow-up 1), and/or early termination.
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: PF-07304814 500 mg 120-hours Continuous Infusion | Part 2: PF-07304814 250 mg 120-hours Continuous Infusion
Number analyzed (Participants) | 6 | 7
ng/mL
  Cmax of PF-07304814: number analyzed (Participants) | 5 | 7
  Cmax of PF-07304814 | 345.3 (70) | 272.6 (281)
  Cmax of PF-00835231 | 2382 (36) | 1265 (20)

24. Secondary Outcome: PF-07304814 (Prodrug) and PF-00835231 (Active Moiety) Plasma PK Parameters: t½ - Part 2: MAD
Description: t½ was defined as terminal half-life. Blood sample collection at approximately within 30 minutes before end of infusion (~120 hours), and at 2 and 6 hours post the end of the infusion, which correspond to approximately 122h and 126h post the start of infusion.
Time Frame: Pre-dose on Day1; Day 2, 3, 5 and 6 (end of treatment day), 7 (Follow-up 1), and/or early termination.
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part 2: PF-07304814 500 mg 120-hours Continuous Infusion | Part 2: PF-07304814 250 mg 120-hours Continuous Infusion
Number analyzed (Participants) | 6 | 7
hour
  t½ of PF-07304814: number analyzed (Participants) | 0 | 0
  t½ of PF-00835231: number analyzed (Participants) | 1 | 3
  t½ of PF-00835231 | 1.79 (NA) — Standard deviation was not applicable because only 1 participant was analyzed. | 2.317 (0.96547)

25. Secondary Outcome: PF-07304814 (Prodrug) and PF-00835231 (Active Moiety) Plasma PK Parameters: Concentration at Steady State (Css) - Part 2: MAD
Description: Css was defined as concentration at steady state. Blood sample collection at approximately 2 and 6 hours post the end of the infusion, which correspond to approximately 122 hours and 126 hours post the start of infusion.
Time Frame: Pre-dose on Day1; Day 2, 3, 5 and 6 (end of treatment day), 7 (Follow-up 1), and/or early termination.
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: PF-07304814 500 mg 120-hours Continuous Infusion | Part 2: PF-07304814 250 mg 120-hours Continuous Infusion
Number analyzed (Participants) | 6 | 7
ng/mL
  Css of PF-07304814: number analyzed (Participants) | 5 | 7
  Css of PF-07304814 | 229.2 (61) | 102.2 (35)
  Css of PF-00835231 | 1720 (44) | 970.2 (16)

ADVERSE EVENTS:
Time Frame: From pre-dose on Day 1 up to 41 days
Description: The same event may appear as both an AE and an SAE. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Part 1: PF-07304814 500 mg 24-hours Continuous Infusion | Part 1: PF-07304814 250 mg 24-hours Continuous Infusion | Part 1: 500 mg Placebo 24-hours Continuous Infusion | Part 1: 250 mg Placebo 24-hours Continuous Infusion | Part 2: PF-07304814 500 mg 120-hours Continuous Infusion | Part 2: PF-07304814 250 mg 120-hours Continuous Infusion | Part 2: Placebo 120-hours Continuous Infusion
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2 | 0/6 | 0/7 | 1/4
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/2 | 1/2 | 1/2 | 1/6 | 2/7 | 1/4
Other Adverse Events (participants affected / at risk) | 1/2 | 1/2 | 2/2 | 2/2 | 2/6 | 3/7 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: PF-07304814 500 mg 24-hours Continuous Infusion (N=2) | Part 1: PF-07304814 250 mg 24-hours Continuous Infusion (N=2) | Part 1: 500 mg Placebo 24-hours Continuous Infusion (N=2) | Part 1: 250 mg Placebo 24-hours Continuous Infusion (N=2) | Part 2: PF-07304814 500 mg 120-hours Continuous Infusion (N=6) | Part 2: PF-07304814 250 mg 120-hours Continuous Infusion (N=7) | Part 2: Placebo 120-hours Continuous Infusion (N=4)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: PF-07304814 500 mg 24-hours Continuous Infusion (N=2) | Part 1: PF-07304814 250 mg 24-hours Continuous Infusion (N=2) | Part 1: 500 mg Placebo 24-hours Continuous Infusion (N=2) | Part 1: 250 mg Placebo 24-hours Continuous Infusion (N=2) | Part 2: PF-07304814 500 mg 120-hours Continuous Infusion (N=6) | Part 2: PF-07304814 250 mg 120-hours Continuous Infusion (N=7) | Part 2: Placebo 120-hours Continuous Infusion (N=4)
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stoma site cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematocrit decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/67/NCT04535167/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/67/NCT04535167/SAP_001.pdf